CLINICAL TRIAL: NCT06364384
Title: Radical Concurrent Chemoradiotherapy With DDP/5-FU and PD-1 Antibody for Newly Diagnosed Non-metastatic Rectal Squamous Cell Carcinoma: A Multicenter, Prospective, Single Arm, Phase II Study(RICH).
Brief Title: Radical Concurrent Chemoradiotherapy With DDP/5-FU and PD-1 Antibody for Non-metastatic Rectal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2024074
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Rectal Squamous Cell Carcinoma
Keywords: PD-1; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 + CRT (Experimental): Patients from experimental group are underwent treatment together with PD-1 monoclonal antibody and radical CRT
  Interventions: Combination Product: PD-1 and CRT

INTERVENTIONS:
Combination Product: PD-1 and CRT — Chemotherapy (/4W): a)DDP 75 mg/m2, d1, intravenous infusion; b)5-FU 1000 mg/m2, d1-4, continuous pumping intravenously; Immunotherapy (/4W): PD-1 monoclonal antibody(sintlimab) 200mg, d1, intravenous infusion; Radiotherapy (at 2rd week after firstime of chemotherapy):Daily single dose of 2Gy, with a total dose of 50-54Gy(clinical I-II stage)/54-59Gy(clinical III stage).

SUMMARY:
The goal of this clinical trial is to learn if PD-1 monoclonal antibody combined with radical chemoradiotherapy works to treat rectal squamous cell carcinoma (rSCC). lt will also learn about the safety of the regime. The main questions it aims to answer are:

Does PD-1 monoclonal antibody combined with radical chemoradiotherapy improve survival prognosis? What is the complete response rate (CCR) of the regime？ Researchers will compare PD-1 monoclonal antibody combined with radical chemoradiotherapy to previous study to see if this regime works to treat rSCCs.

Participants will receive chemotherapy with DDP and 5-FU, immunotherapy with PD-1 monoclonal antibody and radiotherapy with a total dose of 50-54GY.

DETAILED DESCRIPTION:
Rectal squamous cell cancer (rSCC) is a rare malignancy, and its incidence is increasing year by year. Due to the rarity of rSCC, there is no consensus on its epidemiology, pathogenesis, prognosis and treatment management. Due to the limitation of clinical data, there is an urgent need for further clinical exploration and research.

In recent years, the combination of CRT and immunotherapy has attracted more and more attention, as they may have more advantages over CRT alone.A number of prospective clinical trials of PD-1 monoclonal antibody combined with CRT for the first-line treatment of advanced aSCC are also underway (NCT03233711, NCT04230759, NCT05661188, NCT05374252, etc.). Similarly, the efficacy and safety of PD-1 monoclonal antibody in rSCC patients are also worthy of further discussion, in order to further improve the survival prognosis of rSCC patients. Our previous study data showed that the 3-year OS and DFS of radical CRT were 88.9% and 66.7%, respectively, for non-metastatic rSCC, and 100% and DFS for radical CRT combined with immunotherapy, respectively, and CRT combined with immunotherapy significantly improved survival compared with radical CRT (P=0.02).

The goal of this clinical trial is to learn if PD-1 monoclonal antibody combined with radical chemoradiotherapy works to treat rectal squamous cell carcinoma (rSCC). lt will also learn about the safety of the regime. Therefore, we plan to conduct a multicenter, prospective, single-arm, phase II study to provide evidence-based medical evidence for the treatment of locally advanced rectal squamous cell carcinoma.

The primary outcome is 1-year tumor-free survival (DFS), and the secondary outcomes are including 1-year overall survival (OS), 1-year relapse-free survival (RFS), 1-year metastasis free survival (DMFS), 1-year stoma-free survival, incidence of chemotherapy and immunotherapy-related adverse reactions and complete response rate (CRR).

Participants will receive interventions below:

Chemotherapy (/4W): a)DDP 75 mg/m2, d1, intravenous infusion; b)5-FU 1000 mg/m2, d1-4, continuous pumping intravenously; Immunotherapy (/4W): PD-1 monoclonal antibody(sintlimab) 200mg, d1, intravenous infusion; Radiotherapy (at 2rd week after firstime of chemotherapy):Daily single dose of 2Gy, with a total dose of 50-54Gy(clinical I-II stage)/54-59Gy(clinical III stage).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent;
2. 18-75 years old;
3. Patients with pathologically confirmed rectal squamous cell carcinoma;
4. imaging to rule out distant metastases;
5. Peripheral blood and liver and kidney function before treatment within the following allowable limits (tested within 14 days before the start of treatment)

   1. White blood cell (WBC) ≥ 3.0×109/L or neutrophil (ANC) ≥1.5×109/L;
   2. Hemoglobin (HGB) ≥80 g/L;
   3. Platelets (PLT) ≥ 100×109/L;
   4. Hepatic transaminases (AST/ALT) < 3.0 times the upper limit of the normal range;
   5. Total bilirubin (TBIL) < 1.5 times the upper limit of the normal range;
   6. Creatinine (CREAT) < 1.5 times the upper limit of the normal range.
6. ECOG performance status score of 0-2;
7. No history of other malignant tumors in the past.

Exclusion Criteria:

1. Non-treatment-naïve patients who have previously received chemotherapy, radiotherapy or complete surgical resection of rectal squamous cell carcinoma;
2. Distant metastases (M1) confirmed by whole-body CT, MR, or PET-CT (including at least the chest, abdomen, and pelvis);
3. Previous or concurrent presence of other active malignancies (except for malignant tumors that have received curative therapy and have been disease-free for more than 3 years or carcinoma in situ that can be cured by adequate treatment);
4. Major surgery such as laparotomy, thoracotomy, resection of organs by laparoscopic surgery or severe trauma within the past 4 weeks (the surgical incision should be completely healed before randomization);
5. Active coronary artery disease, severe/unstable angina pectoris or newly diagnosed angina pectoris or myocardial infarction within 12 months prior to enrollment in the study;
6. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis within the past 6 months;
7. New York Heart Association (NYHA) Class II or above congestive heart failure;
8. Prior receipt of any investigational drug;
9. Pregnant or lactating women;
10. Any medical condition that is unstable or would affect patient safety and their compliance with the study;
11. Patients judged by the investigator to be unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
3-year tumor-free survival(DFS) | 3 year
  The proportion of patients who do not have any of the following events from the beginning of randomization to the end of the first year

SECONDARY OUTCOMES:
1-year overall survival (OS) | 1 year
  Time interval from the date of randomization to death
1-year relapse-free survival (RFS) | 1 year
  Time interval from the date of randomization to the onset of recurrence
1-year metastasis free survival (DMFS) | 1 year
  Time interval from the date of randomization to the occurrence of distant metastases
Incidence of chemotherapy and immunotherapy-related adverse reactions | through study completion, an average of 6 months
  The occurrence of chemotherapy and immune-related side effects during treatment
Complete response rate (CRR) | through study completion, an average of 6 months
  The proportion of the total number of patients with complete response after treatment to the total number of evaluable cases in solid tumor treatment studies
1-year stoma-free survival | 1 year
  The occurrence of stoma

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China